CLINICAL TRIAL: NCT00885911
Title: Evaluation of the Intubating Laryngeal Airway in Children - Phase 1
Brief Title: Evaluation of the Intubating Laryngeal Airway in Children
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Simon Whyte, Principle Investigator, University of British Columbia
Other Study IDs: H08-01196
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Intubating Laryngeal Airway
Keywords: Intubating laryngeal airway; pediatric; observational study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Extraglottic device: The laryngeal mask airway (LMA) used during pediatric anesthesia for routine and difficult airway management.

SUMMARY:
The Air-Q® intubating laryngeal airway (Air-Q® ILA) is an extraglottic device specifically engineered for use both as a stand-alone laryngeal mask airway (LMA) and as a rescue device or "Plan B" device in the event of a difficult airway. As with some other types of LMA, it is then possible to insert an endotracheal tube (ETT) through the Air-Q® ILA, either blindly or mounted on a fibreoptic bronchoscope (FOB), to achieve endotracheal intubation. This will be a prospective observational study of the Air-Q® ILA's performance.

DETAILED DESCRIPTION:
Hypothesis: The Air-Q® intubating laryngeal airway (Air-Q® ILA) will: (1) perform satisfactorily as a primary airway; (2) perform comparably or better than the ProSeal™ LMA (PLMA); and (3) act as an excellent conduit for fibreoptic intubation.

Background: The laryngeal mask airway (LMA) is used during pediatric anesthesia for routine and difficult airway management. The ideal pediatric LMA device would provide excellent sealing at low pressure; facilitate easy endotracheal intubation; and be available in pediatric sizes. Such a device would be an invaluable addition to difficult pediatric airway management plans and, by increasing the likelihood of quickly and effectively securing the difficult airway, and decreasing the risk of catastrophic hypoxemia, would increase perioperative safety for children. The Air-Q® ILA is a modified LMA device whose features encompass the characteristics of the ideal LMA. Our objective is to determine whether or not this new airway device is an improvement over the current standard of care.

Specific Objectives:

1. To test the performance characteristics of the Air-Q® ILA as a primary airway in clinical pediatric anesthetic practice;
2. To compare Air-Q® ILA performance to the current best option, the PLMA for sizes 1.0, 1.5, 2.0 and 2.5; To evaluate the performance characteristics of the Air-Q® ILA as a conduit for fibreoptic intubation

Methods:

Recruitment of subjects: With ethical and institutional review board approval, and with written parental informed consent, we will recruit children, ages 0-12 years, undergoing elective surgery. Children with ASA status IV-V, abnormal or contraindicated cervical spine flexion/extension/rotation, contraindication to LMA placement, or requiring emergency surgery will be excluded. All children will undergo intravenous induction of anesthesia, as per our routine institutional practice.

Administration of Air-Q® ILA: In phase 1, the age/weight-appropriate Air-Q® ILA will be inserted in each child and assessed, using published, objective criteria. In phase 2, either a PLMA or an Air-Q® ILA will be inserted and assessed. The first LMA will then be removed and the other device inserted and assessed. The order of insertion will be determined by block randomization. In phase 3, the Air-Q® ILA will be inserted and, after ensuring adequate ventilation, a study investigator will undertake fibreoptic-guided endotracheal intubation through the Air-Q® ILA, after which the Air-Q® ILA will be removed. The performance characteristics of the Air-Q® ILA as a conduit for fibreoptic-guided endotracheal intubation will be evaluated.

Data analysis: Phase 1 will generate descriptive data on several validated performance characteristics. The primary outcome measure will be the oropharyngeal leak pressure (OLP) value. In phase 2, we will compare OLP values using paired t- tests. We will conduct appropriate statistical analysis of the data on the other assessment variables, which are all secondary outcome measures. In phase 3, the arterial oxygen saturation, heart rate, and rise in end-tidal CO2 will be reported as outcome variables, along with the time taken to complete the fibreoptic intubation. Descriptive data will be presented as mean ± SD, median (range), counts (percentages or proportions) as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Ideal body weight as determined from weight/height centile curves (> 3rd & < 97th centiles)
* Elective surgery
* Appropriate subject and procedure for airway management by LMA

Exclusion Criteria:

* ASA status IV-V
* Emergency surgery
* Abnormal or contraindicated cervical spine flexion/extension/rotation
* Contraindication to LMA placement:

  * Aspiration risk; gastro-oesophageal reflux disease
  * Clinically significant pulmonary disease
  * Coagulopathy
  * Distorted airway anatomy judged likely to compromise LMA placement
  * Allergy to any LMA components

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Perioperative safety for children. A device that would be an invaluable addition to difficult pediatric airway management plans, increasing the likelihood of quickly and effectively securing the difficult airway, and decreasing the risk of catastrophic hypoxemia.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2009-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Whyte, MD, Principal Investigator — University of British Columbia; Stephan Malherbe, MD, Study Director — University of British Columbia; Andrew Morrison, MD, Study Director — University of British Columbia
Locations (1):
- British Columbia Children's Hospital Department of Anesthesia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Whyte SD, Cooke E, Malherbe S. Usability and performance characteristics of the pediatric air-Q(R) intubating laryngeal airway. Can J Anaesth. 2013 Jun;60(6):557-63. doi: 10.1007/s12630-013-9918-6. Epub 2013 Mar 22. PMID 23519724